CLINICAL TRIAL: NCT01878357
Title: Impact of Mass Screening and Selective Treatment With Dihydroartemisinin-piperaquine Plus Primaquine on Malaria Transmission in High Endemic Area, Belu Regency, Nusa Tenggara Timur Province, Indonesia: a Randomized Cluster Trial
Brief Title: Surveillance and Treatment With Dihydroartemisinin-piperaquine Plus Primaquine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Inge Sutanto, Prof. DR. dr., Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTC Belu
Record Dates: First submitted 2013-06-04; First posted 2013-06-14 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Malaria
Keywords: MST; Malaria; Indonesia; Transmission
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DHP monthly (Experimental): Three mass screening and selective treatment using dihydroartemisinin-piperaquine and primaquine i.e. on month 1 (MST1), month 2 (MST2), and month 3 (MST3) with an interval of 6 weeks between each MST
  Interventions: Drug: dihydroartemisinin-piperaquine; Drug: primaquine
- DHP bi-monthly (Experimental): Two mass screenings and selective treatment using dihydroartemisinin-piperaquine and primaquine i.e. on month 1 (MST1) and month 3 (MST3) with an interval of 3 months.
  Interventions: Drug: dihydroartemisinin-piperaquine; Drug: primaquine
- Arm 3 (No Intervention): Without MST

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — Treatment will be given to all malaria-positive individuals on microscopic examination. The dosage will be calculated based on body weight. The drug that will be given is 3-day dihydroartemisinin-piperaquine (DHP) treatment. The drug will be given by health care personnel at their houses assisted by health care volunteers of the integrated health post (Posyandu cadre).
  Other Names: D-artepp
  Arms: DHP bi-monthly; DHP monthly
Drug: primaquine — One day primaquine (PQ) treatment will be given for P. falciparum infected subjects. For patients who are infected by P. vivax and P. ovale,PQ will be given for 14 days
  Other Names: PQ
  Arms: DHP bi-monthly; DHP monthly

SUMMARY:
Mass Drug Administration (MDA) and Mass Screening and Selective Treatment (MST) might be applied as strategies for eliminating malaria when focusing on transmission stages. Many studies either with MDA or MST has been done in low transmission areas demonstrated the impact of those activities to reduce malaria transmission. However, in high transmission such study is still very limited which is becoming the reason behind this study.

A randomized cluster trial of MST study using dihydroartemisinin-piperaquine plus primaquine (DHP + PQ) will be conducted in some villages at the Belu regency, Nusa Tenggara TImur province, Central Indonesia. There will be three arms in the study, i.e. (1) intervention arm of mass screening and treatment with interval of 6 weeks; (2) intervention arm of mass screening and treatment with interval of 3 months and (3) control arm without mass screening and treatment. The intervention arm with 6 weeks interval represents a new proposed method to detection malaria infections, while the intervention arm with 3 month interval represents the Ministry of Health current policy of active case detection in Indonesia, and the third arm will serve as the control for Ministry of Health's policy.

The study will be conducted in 6 months period and evaluate various parameters including malaria incidence and proportion of anemia in monthly cohort school children (in arm1, 2 and 3), in addition to malaria prevalence in the community (only in arm 1 and arm 2). All positive subject in all arms will receive supervised treatment. Secondary objectives are the proportion of gametocytemia in the community, the proportion of malaria antibody of various age groups, population genetic of local parasite, submicroscopic incidence based polymerase chain reaction and the proportion of infective mosquitoes. Data analysis will be performed according to the method for cluster randomized trial evaluation.

DETAILED DESCRIPTION:
Study Site

The study will be conducted at Belu regency (south latitude 90 - 100; east longitude 1240- 1260) which located in the Nusa Tenggara Timur province, central part of Indonesia.

Atambua District Health Office reported that most of high endemic malaria areas were situated in the southern part of the regency in 2011. The highest Annual Parasite Incidence (API) reported was in the subdistrict of Wewiku (72.1 cases/1,000 people). Therefore, this study will focus in high case incidence of villages in Wewiku sub-districts.

Study design overview and demographic census

The study design is "randomized cluster trial" by microscopic malaria screening at high malaria incidence at village level. Two-four villages with malaria prevalence of >8% or sub-villages with malaria prevalence > 10% in school children will be selected as study villages or sub-villages.

Census visit will be performed in all target villages. All clusters will be then listed and randomized to one of study arm using generated randomization softwares.

There will be 3 study arms, i.e. (1) 6 weeks interval of MST, (2) 3 months interval of MST; and (3) control without MST. Each MST should cover at least 80% of the villagers.

Treatment will be given to all malaria-positive individuals on microscopic examination. The treatment will be provided based on suitable dose for body weight as recommended by the Ministry of Health, Republic of Indonesia (Table 1). The drug that will be given is 3-day dihydroartemisinin-piperaquine (DHP) treatment and 1-day primaquine (PQ) treatment for P. falciparum. For patients who are infected by P. vivax and P. ovale,PQ will be given for 14 days; while the dose of DHP is equal to the dose for P. falciparum infection. Treatment for P.malariae infected subjects is similar with that for P. falciparum but without PQ. For individuals in all arms, the drug will be given by health care personnel at their houses assisted by health care volunteers of the integrated health post (Posyandu cadre).

Ethics Consideration

An informed consent will be collected from every head of families or their representative. They have 1 week to consider whether they will participate in our study or not.

Adverse events will be identified and recorded in Case Report Form by field team in collaboration with cadres and primary health center attendants. These subjects will be given symptomatic treatment at the village/sub-village level or at the local health center. Relationship between adverse event and study drug will be determined by Data Safety and Monitoring Board (Prof Rianto Setiabudy, dr Erni Juwita Nelwan and dr Hasan Basri) who will also decide how often the data will be sent to Jakarta. Specific Adverse Event are black urine, gastro intestinal disturbances, blue lips and breathless.

Serious Adverse events is an adverse event which becomes serious and could endanger the life of subjects, cause prolonged hospitalization and disability to conduct normal life. The Data Safety and Monitoring Board will be recorded in Severe Adverse Event form and reported to Principal Investigator, sponsors, Ethic Committee, Regulatory and Data Safety and Monitoring Board within 24 hours. Severe Adverse Event subjects will be treated in Atambua Hospital until recover completely. All expenses will be paid by sponsor. Complete Severe Adverse Event report will be distributed within one month after the occurrence of Severe Adverse Event.

Evaluation Malaria incidence Inclusion Criteria Children at elementary school (6-12 year old) of the all selected clusters despite of random allocation.

Sample size Sample size is calculated based on the differences of malaria incidence between before and after intervention in each arm. Baseline incidence is determined from positive-malaria children in monthly cohort between MST1 and MST3 in arm 1 or MST1 until MST3 in arm 2. Malaria incidence in the arm 2 is assumed to remains constant at 0.7 new cases/person-year during study(unpublished data). The impact of the intervention arm is expected to reduce malaria incidence maximum by 50% to 0.35 new cases/person-year. With the proposed sample size of 70 children per arm, we will have a power of 82% to detect a significant difference. Considering a 10% of loss to follow-up and a design effect of cluster-randomized trial 1.5, we will recruit 115 children per arm.

All school-age children who participate in the study and have malaria-positive blood smears will receive complete treatment as previously mentioned. The antimalaria drug will be given by direct observation treatment (DOT) technique or under supervision performed by school teachers with the assistance of the health care volunteers.

Blood samples drawn by pricking the finger tip in school-age children are used for microscopic examination, Polymerase Chain Reaction assay, hemoglobin measurement, serological examination for malaria antibody and Glucose-6-Phosphate Dehydrogenase deficiency assessment.

Anemia in malaria infection

Inclusion criteria Elementary school children aged 6-12 years who participate in cohort study.

Sample size Sample size calculation is performed by WinPepi software with the assumed anemia proportion of 25% and 50% in arm 1 and arm 2, respectively (5% significance level, 80% power, and 1:1 sample size ratio). Required sample size would be 58 school-age children per arm. We will recruit115 school children after considering design effect of 1.5,and drop out level of 10% and sample size for malaria incidence

Blood samples are drawn by pricking the finger tip of the elementary school children using microtainer as much as 0.25 ml. Simultaneously, the thick and thin blood smears are made for microscopic examination of malaria and hemoglobin level measurement. The collected blood samples in the tube containers are delivered to the laboratory for distribution of above mentioned assays.

Malaria prevalence

Inclusion criteria All villagers of the selected clusters ( arm 1: MST1, 2, 3 and arm 2: MST1, MST3), except elementary school children who participated in cohort study. Cluster chosen should be located in villages with endemicity of more than 8% or sub-villages of more than 10%.

Sample size Sample size is calculated based on the differences of malaria prevalence before and after treatment in the arm 1 and arm2. The malaria prevalence used in the study is 15%, which is expected to decrease by 30% in arm 1 and persistent in arm 2. Sample size calculation is performed by WinPepi software with the assumed probability proportion of 10% and 15% in arm 1 and arm 2, respectively (5% significance level, 80% power, and 1:1 sample size ratio). Required sample size would be 686 subjects. We will recruit 1029 subject after considering design effect of 1.5.

All villagers participated in both arms who have malaria-positive blood smears will be treated completely as previously described. The antimalaria drug will be given by direct observation treatment (DOT) technique or under supervision performed by health care personnel with the assistance of the health care volunteers to ensure that the treatment coverage would reach 100%.

Blood samples are drawn by pricking the finger tip of the individuals in the community using microtainer as much as 0.25 ml for > 1 year-old children and adults or 0.1 ml for infants (the blood samples are drawn by pricking the finger tip of their toes). Simultaneously, the thick and thin blood smears are made for microscopic examination of malaria.

The change of malaria antibody in population

Inclusion criteria All villagers of the selected clusters ( arm 1: MST1 & 3 and arm 2: MST1 &3) and children enrolled in cohort study from all arms.

Sample size Sample size is calculated based on the proportion of altered malaria antibody before and after intervention in arm 1 and arm 2. The seropositive prevalence rate used in the study is 50% (unpublished data), which is expected to be seronegative as much as 25% in arm 1; while the change in the arm 2 would be 10%. Sample size calculation is performed by WinPepi software assuming that the proportion of seroconversion (from + to -) is 25% in arm 1 and 10% in arm 2 (5% significance level, 80% power, and 1:1 sample size ratio). Required sample size would be 321 subjects. After considering design effect of 1.5, we will recruit 482 subjects per arm and this will be randomized from community blood collected sample.

Gametocyte carriage in the population

Inclusion criteria All villagers of the selected clusters ( arm 1: MST1, 2, 3 and arm 2: MST 1 &3) but not included elementary school children who participated in cohort study.

Sample size Sample size is calculated based on the proportion of gametocyte carriages before and after intervention in both arm.The assumption of gametocyte proportion rate used in the study is 20%, which is expected to decrease by 40% in arm 1 and decrease by 10% in the arm 2. Sample size calculation is performed by WinPepi software by assuming that the reduced proportion of gametocyte carriage of 40% in arm 1 and 10% in arm 2 (5% significance level, 80% power, and 1:1 sample size ratio). Required sample size would be 338subjects. After considering design effect of 1.5, we will recruit 507 subjects per arm that will be randomized from 1029 community participants

Incidence based on molecular characterization

Inclusion criteria All children in cohort study (arm 1 and 2).

Sample size Blood samples are taken from all school-age children enrolled in cohort study or children per arm.

Oocyst and sporozoite rate in vector mosquitoes Oocyst and sporozoite rate in mosquitoes will be determined at three points: baseline, week 6, and month 3. Mosquitoes will be collected within a week before nearest MST carried out. All collected mosquitoes in the period of study as mentioned before will be subjected to the laboratory examination.

Parasite population genetic

Inclusion criteria:

Fifty samples for any malaria species (positive P. falciparum and P. vivax) at every mass blood survey from each arm (arm 1 and arm 2). This number is considered representative of local parasite genetic.

ELIGIBILITY:
Inclusion Criteria:

* All villagers of the all selected clusters

Exclusion Criteria:

* Pregnant women during their first trimester
* Single dose primaquine should not be given for infants less than 1 year-old, pregnant women in all trimesters of pregnancy, breast-feeding mother and patients with G6PD deficiency

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1488 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Malaria incidence | 6 months
  Malaria incidence in children at the elementary schools (all arms)

SECONDARY OUTCOMES:
Anemia | 6 months
  Proportion of anemia in elementary school children (all arms)

OTHER OUTCOMES:
Malaria prevalence | 3 months
  Malaria prevalence in all age groups (only arm 1 and arm 2)
Antimalaria antibody | 6 months
  Seroconversion rate of antimalaria antibody in all age groups (all arms)
Infective vector | 3 months
  Oocyte and sporozoite rates in vector mosquitoes (all arms)
Gametocyte carriage | 3 months
  Gametocyte carriage rate in all age groups (arm 1 and arm 2)
Parasite genetic diversity | 3 months
  Genetic diversity of Plasmodium falciparum and P. vivax(arm 1 and arm 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Kecamatan Wewiku, Betun, East Nusa Tenggara, Indonesia

REFERENCES:
- [Background] Shekalaghe SA, Drakeley C, van den Bosch S, ter Braak R, van den Bijllaardt W, Mwanziva C, Semvua S, Masokoto A, Mosha F, Teelen K, Hermsen R, Okell L, Gosling R, Sauerwein R, Bousema T. A cluster-randomized trial of mass drug administration with a gametocytocidal drug combination to interrupt malaria transmission in a low endemic area in Tanzania. Malar J. 2011 Aug 24;10:247. doi: 10.1186/1475-2875-10-247. PMID 21864343
- [Derived] Kosasih A, Koepfli C, Dahlan MS, Hawley WA, Baird JK, Mueller I, Lobo NF, Sutanto I. Gametocyte carriage of Plasmodium falciparum (pfs25) and Plasmodium vivax (pvs25) during mass screening and treatment in West Timor, Indonesia: a longitudinal prospective study. Malar J. 2021 Apr 9;20(1):177. doi: 10.1186/s12936-021-03709-y. PMID 33836772
- [Derived] Sutanto I, Kosasih A, Elyazar IRF, Simanjuntak DR, Larasati TA, Dahlan MS, Wahid I, Mueller I, Koepfli C, Kusriastuti R, Surya A, Laihad FJ, Hawley WA, Collins FH, Baird JK, Lobo NF. Negligible Impact of Mass Screening and Treatment on Mesoendemic Malaria Transmission at West Timor in Eastern Indonesia: A Cluster-Randomized Trial. Clin Infect Dis. 2018 Oct 15;67(9):1364-1372. doi: 10.1093/cid/ciy231. PMID 29579195